CLINICAL TRIAL: NCT00557596
Title: A Phase 1-2, Multicenter, Open-Label Study of The X-Linked Inhibitor of Apoptosis (XIAP) Antisense AEG35156 Given in Combination With Gemcitabine in Patients With Advanced Pancreatic Cancer
Brief Title: A Phase 1-2, XIAP Antisense AEG35156 With Gemcitabine in Patients With Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aegera Therapeutics (Industry)
Responsible Party: Jacques Jolivet, MD, Senior VP Clinical, Aegera Therapeutics Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEG35156-201
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Carcinoma; Pancreas
Keywords: Pancreatic; antisense; oligonucleotide; gemcitabine
MeSH Terms: conditions — Carcinoma | interventions — AEG 35156

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AEG35156 — AEG35156 will be given as a 2-hour intravenous infusion once weekly, only on weeks when gemcitabine is administered, with a 2-hour loading dose given daily in the 2 days immediately prior to Day 1 (on Days -2 and -1) only in Cycle 1

SUMMARY:
This is an open-label multicenter, phase 1-2 study. Following determination of the recommended AEG35156 dose in combination with gemcitabine in the initial Phase 1 part of this study, additional patients will be enrolled in the Phase 2 part of the study to assess the activity of the combination first-line in advanced pancreatic cancer.

DETAILED DESCRIPTION:
Apoptotic induction in cancer cells is a sought after therapeutic goal. Most successful anticancer agents activate apoptosis pathways in the cancers they treat. Apoptotic pathways in cells appear to converge on a single family of enzymes, the caspases, which are proteases that dismantle the cell in an orderly, non-inflammatory fashion, resulting in cell death. The X-linked Inhibitor of Apoptosis (XIAP) is the only known cellular inhibitor of caspases, its over expression thereby blocks the principal means of apoptosis. A wide range of evidence indicates that cellular overexpression of members of the IAP family is a fundamental means by which many cancer cells evade death, even in the presence of strong extrinsic (death receptor-mediated) and intrinsic (mitochondria-mediated) apoptotic cues. The inhibition of cellular XIAP activity, specifically in cancer cells under stress and primed for apoptosis by chemotherapeutic agents, is viewed as a powerful means of tipping the balance towards cell death. In particular, XIAP has been shown to be overexpressed in pancreatic cancer and to play an important role in gemcitabine resistance. AEG35156 is a second generation antisense which targets XIAP mRNA to lower XIAP levels and the apoptotic threshold of cancer cells, enhancing their sensitivity to intrinsic death and chemotherapy. AEG35156 may thus enhance the anticancer activity of gemcitabine in patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed advanced pancreatic adenocarcinoma who are candidates for first-line gemcitabine therapy
* Karnofsky performance >70%
* One or more metastatic tumors measurable by RECIST criteria on CT scan or MRI (Phase 2 part only)
* Life expectancy of at least 3 months
* Age > 18 years
* Signed, written IRB-approved informed consent
* A negative serum pregnancy test (if applicable)
* Acceptable liver function:
* Bilirubin < 1.5 times the institution's upper limit of normal
* AST (SGOT), ALT (SGPT) and Alkaline phosphatase < 2.5 times the institution's upper limit of normal
* Acceptable renal function:
* Serum creatinine within normal limits, OR calculated creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Acceptable hematologic status:
* Granulocyte > 1500 cells/uL
* Platelet count > 100,000 plt/uL
* Hemoglobin > 9.0 g/dL
* Acceptable coagulation status:
* PT within normal limits
* PTT within normal limits
* For women of child-producing potential, the use of effective contraceptive methods during the study
* Prior radiotherapy for local disease is allowed provided disease progression has been documented, and treatment completed at least 4 weeks prior to registration

Exclusion Criteria:

* Prior chemotherapy for pancreatic cancer, except for 5-fluorouracil or gemcitabine given as a radiosensitizer
* Active progressive brain metastases including the presence of any related symptoms or need for corticosteroids. A CT or MRI scan of the head is necessary in patients with a history of brain metastases to document the stability of prior lesions.
* Known bleeding diathesis or concurrent treatment with anticoagulants except patients on non-therapeutic line maintenance coumadin
* Pregnant or nursing women. NOTE: Women of child-bearing potential must agree to use adequate contraception (sterile or surgically sterile; hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Men who are unwilling to use acceptable forms of birth control when engaging in sexual contact with women of child bearing potential
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Known infection with HIV, hepatitis B, or hepatitis C
* Serious nonmalignant disease that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
* Patients who are currently receiving any other investigational agent. Subjects who have used a previous antisense oligonucleotide in the last 90 days will be excluded
* Unwillingness or inability to comply with procedures required in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
To determine the recommended dose of AEG35156 when used in combination with gemcitabine and the change in response rate of gemcitabine in patients | 1 year

SECONDARY OUTCOMES:
To determine progression-free survival. | 2 years
To establish the pharmacokinetics of AEG35156 and gemcitabine when used in combination. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D Von Hoff, MD, FACP, Principal Investigator — TGen Clinical Research Services at Scottsdale Healthcare; Jacques Jolivet, MD, FACP, Study Director — Aegera Therapeutics, Inc.
Locations (4):
- United States (4):
  - Scottsdale Healthcare - SHEA, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Arizona Cancer Center - University of Arizona, Tucson, Arizona
  - Gabrail Cancer Center, Canton, Ohio